CLINICAL TRIAL: NCT03231891
Title: Inherited CAncer REgistry (ICARE) Initiative
Brief Title: Inherited CAncer REgistry
Acronym: ICARE
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Responsible Party: Principal Investigator, Tuya Pal, Associate Director for Cancer Health Disparities, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC MD 1712
Record Dates: First submitted 2017-07-24; First posted 2017-07-27 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 100 Years
Biospecimen Retention: Samples With DNA — Collection of blood, saliva/cheek swab, urine, and/or other biological specimens may be requested from participants. Tissues saved during previous surgeries as part of the patient's treatment may be requested.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the Inherited CAncer REgistry (ICARE) Initiative is to provide individuals interested in participating in studies focused on inherited cancer predisposition the opportunity to enroll in a research registry. Efforts through the registry include, but are not limited to, contribution of data to observational studies, targeted gene-specific studies, and education and outreach efforts for both participants and recruiting healthcare providers. Participants are given the opportunity to learn about and participate in other efforts for which they may be eligible.

All participants and recruiting healthcare providers receive educational newsletters twice per year which contain research and clinical updates in the field of cancer genetics. Providers who recruit patients can also access monthly web-based genetics case conferences which focus on different topics each month and are generally attended by a guest expert who provides background information on the topic as well as comments on the case presentations.

Participation in ICARE involves completion of an informed consent form, baseline questionnaire, follow-up questionnaires every two years, and medical record/tumor releases, as applicable. There is no cost to participate and all correspondence can be facilitated through phone, email, or mail.

Enrollment can be completed either through a traditional paper-based consenting method (i.e. postal mail) or through the online enrollment option available on the ICARE website (InheritedCancer.net). If you are a patient interested in learning more or a provider interested in recruiting to ICARE, please visit our website where you may complete an online contact form requesting a study team member contact you.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Able and willing to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals interested in participating in inherited cancer research studies.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2017-02-27 (Actual); Primary Completion 2034-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Establish and maintain a registry of individuals who are interested in participating in studies of the genetics of cancer and other related investigations. | Up to 100 years

CONTACTS AND LOCATIONS:
Overall Officials: Tuya Pal, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Inherited Cancer Registry (ICARE) Website — http://inheritedcancer.net